CLINICAL TRIAL: NCT01205347
Title: Phase 4 Study of the Effect of Statin Treatment on Insulin Sensitivity During Myocardial Infarction
Brief Title: Effect of Statin Treatment on Insulin Sensitivity During Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brasilia Heart Study Group (Other)
Responsible Party: Principal Investigator, Andrei C. Sposito, Professor of Cardiology, Brasilia Heart Study Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Statin_InsulinSensitivity
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Myocardial Infarction
Keywords: Statin; Myocardial infarction; Insulin sensitivity
MeSH Terms: conditions — Myocardial Infarction; Insulin Resistance | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin 80mg (Experimental): Simvastatin 80mg once a day
  Interventions: Drug: Simvastatin 80mg
- Simvastatin 10mg (Active Comparator): Simvastatin 10mg once a day
  Interventions: Drug: Simvastatin 10mg

INTERVENTIONS:
Drug: Simvastatin 80mg — Simvastatin 80mg once a day
  Other Names: Zocor
  Arms: Simvastatin 80mg
Drug: Simvastatin 10mg — Simvastatin 10mg once a day
  Other Names: Zocor
  Arms: Simvastatin 10mg

SUMMARY:
Stress hyperglycemia during myocardial infarction (MI) is related to mortality at short and long term. Recent studies, however, revealed that chronic statin treatment may decrease both insulin sensitivity and secretion immediately after statin therapy initiation. This study aim was to investigate the dose-dependent effect of statins on insulin sensitivity in patients in the acute phase of MI.

DETAILED DESCRIPTION:
Stress hyperglycemia during myocardial infarction (MI) is a predictor of worse prognosis at short and long term. From the mechanistic standpoint, hyperglycemia can attenuate thrombolysis, increase platelet aggregation, induce coronary vasoconstriction, reduce oxygen transport and prolong endothelial inflammation after MI. Consistently, observational data indicates that glucose normalization improves survival in hyperglycemic patients hospitalized with MI.

High dose potent statins have been included in the early treatment of acute coronary syndromes (ACS) based upon a broad range of potentially beneficial mechanisms. Recent studies, however, revealed that chronic statin treatment may increase the incidence of type 2 diabetes mellitus in a dose-dependent manner. Moreover, according to studies in cellular and animal models, such decrease in insulin sensitivity may be observed immediately after statin therapy initiation. By inference, one may speculate that statin treatment initiated at the acute phase of MI may potentially favor the appearance or aggravation of stress hyperglycemia. To date, however, this hypothesis has not been investigated. Hence, this study aim was to investigate the dose-dependent effect of statins on insulin sensitivity in patients in the acute phase of MI.

ELIGIBILITY:
Inclusion Criteria:

* Less than 24 hours after the onset of MI symptoms
* ST-segment elevation of a least 1 mm (frontal plane) or 2 mm (horizontal plane) in two contiguous leads
* Myocardial necrosis, as evidenced by increased Creatine Kinase-MB (CK-MB) and troponin levels

Exclusion Criteria:

* Diabetes or prior use of statins in the last 6 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 5 days
  Insulin sensitivity as determined by hyperinsulinemic normoglycemic clamp

SECONDARY OUTCOMES:
Activation of insulin receptor substrate (IRS-1) and Akt protein | 5 days
  Verify the degree of phosphorylation of insulin receptor substrate (IRS-1) and Akt protein estimated by Western Blotting of the abdominal adipose tissue obtained by biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, MD PhD, Study Chair — Faculty of Medical Sciences, State University of Campinas
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil